



# STATISTICAL ANALYSIS PLAN FOR EXPO – PHASE 1

Date: 08/06/2022

Version: 4

Extended-release pharmacotherapy for opioid use disorder (EXPO): Protocol for an open-label randomised controlled trial of injectable maintenance buprenorphine with personalised psychosocial intervention. The EXPO study.

IRAS Project ID: 255522

REC: London - Brighton and Sussex

EudraCT: 2018-004460-63

Based on protocol version: V5.1 (06/10/2021)

**Chief Investigator:** 

Mike Kelleher

Co-Investigators/Co-Applicants

John Marsden

Luke Mitcheson

Caroline Murphy

Joanna Kelly

Eilish Gilvarry

Ed Day

Jonathan Dewhurst

Fiona Cowden

Trial Manager

Jatinder Bisla

Senior Trial Statistician

Zoë Hoare

Trial Statistician

**Rachel Evans** 

**Approval signatures** 

Rachel Evans

Author's Name

Date and Signature

08/06/2022

Zoë Hoare

Second Statistical Advisor

Date and Signature

08/06/2022

Mike Kelleher

Chief Investigator

Date and Signature

8/1/122

**Professor Tim Millar** 

**DMC Chair** 

Date and Signature

Professor Richard Holland

TSC Chair

Date and Signature

10/6/2022

12/1/22

**DOCUMENT HISTORY** 

| cation Ided Ing data added Ing current Ided Ided Ided Ided Ided Ided Ided Ide |
|---|
| ng data added ing current clarified led added, and ences updated ons (ineligible |
| ng data added ing current clarified led added, and ences updated ons (ineligible |
| ng data added ing current clarified led added, and ences updated ions (ineligible |
| clarified<br>led<br>added, and<br>ences updated |
| clarified<br>led<br>added, and<br>ences updated<br>ions (ineligible |
| clarified<br>led<br>added, and<br>ences updated<br>ons (ineligible |
| led added, and ences updated ons (ineligible |
| added, and<br>ences updated<br>ons (ineligible |
| ences updated<br>ons (ineligible |
| ons (ineligible |
| rviews) and |
| or of final visit |
| 8 |
| late |
| er added |
| t study phase |
| ons updated |
| stments for |
| added |
| randomised |
| tocol violation |
| t that missing |
| issing data for |
| me |
| test protocol |
| ing data due to |
| ng days off end |
| e to final visit |

| testing | to 161 to day 0 to 168 |
|---|---|
| analyses or model | Update of grace period sensitivity from day 0 |
| 6.9 Sensitivity | Table 3 dates of UDS collection updated |
| outcome measures | within this SAP |
| calculations of | not be conducted as part of the analysis |
| 5.2 Definitions and | Clarification that objective 3, measure 3 will |
| 6.1 Analysis timeframe | Update to planned analysis timelines |
| Appendix 3 | Addition of MOCA scoring |
| | SURE to align with correct scoring. |
| Appendix 2 | Adjustments to scoring of CEQ-F, WSAS and |
| Section 3.1 | Background text updated to align with latest protocol |
| document | Esp emended to ESP |
| throughout | Bup amended to BUP-SL |
| Acronym table and | Met amended to MET |
| A | XR-Bup amended to BUP-XR |
| | period |
| | Addition of sensitivity analysis for Grace |
| Section 6.9 | administration error. |
| * | addition of 14-day TLFB truncated analysis for |
| | Clarification of per protocol and mITT and |
| | UDS missing data sensitivity analysis, |
| | Updates to sensitivity analysis; Addition of |
| Section 6.8 | Detail on sub group analysis added in |
| Section 6 | Analysis timelines updated |
| Section 5.3 | reported in final analysis report |
| | Update to text to clarify safety data being |
| measures | interviews |
| Section 5.2 other | PHQ-15, PHQ4 and OSTQOL added for exit |
| | notes and rule for where this has occurred |
| | being conducted early) and use of medical |

4

Rachel Evans

4.6 Missing Data

Addition of sentence to clarify item imputation for continuous outcome measures. MOCA removed as potential predictor of missingness as measure was unobtainable during study due to COVID.

Other minor clarifications.

\*Version 1 signed off by Author, Principal Statistician, CI and TSC chair. Updates occurred before DMEC chair final sign off.

# **TABLE OF CONTENTS**

| 1. | Acronyms and definition of terms | 8 |
|----|--------------------------------------------------------|------|
| 2. | Statistical analysis plan authorship | 10 |
| 3. | Introduction | 10 |
| | 3.1 Background and Design | 10 |
| | 3.2 Trial Objectives | 14 |
| | 3.3 CONSORT Diagram | |
| 4. | Statistical Principles | 16 |
| | 4.1 Sample size justification | 16 |
| | 4.2 Randomisation | 16 |
| | 4.3 Levels of confidence and p-values | 17 |
| | 4.4 Adherence | 17 |
| | 4.5 Protocol Violations | 18 |
| | 4.6 Missing Data | 18 |
| | 4.7 Assumption Checking | 20 |
| 5. | Data | 21 |
| | 5.1 Time points of outcomes measures | 22 |
| | 5.2 Definitions and calculations of outcome measures | 24 |
| | 5.3 SAFETY data | . 28 |
| 6. | Statistical analyses | 29 |
| | 6.1 Analysis Time Frame | 29 |
| | 6.2 Baseline Analysis | . 29 |
| | 6.3 Interim Analysis | . 29 |
| | 6.4 CONSORT Analysis | . 29 |
| | 6.5 Descriptive statistics | . 30 |
| | 6.6 Analysis of primary outcome | . 31 |
| | 6.7 Analysis of secondary outcomes | . 31 |
| | 6.8 Subgroup analyses | . 32 |
| | 6.9 Sensitivity analyses or model testing | . 32 |
| | 6.10 Exploratory analyses | . 35 |
| 7. | Software | . 35 |
| | References | |
| Α | ppendices | . 36 |
| | Appendix 1 – Poisson Regression Analysis Decision Tree | |

| Appendix 2 – Objectives and associated outcome measures and characteristics 38 |
|---|
| Appendix 3 - Outcome measures summary and scoring table |
| Appendix 4 – Assumptions of models |
| Table 1: List of outcome measures to be collected and time point of collection 23 |
| Table 2: Planned target timeline for analysis dependent on recruitment period |
| Table 3: Summary of UDS data collection during trial following COVID-19 impacts |
| Figure 1: Randomisation summary for Phase 1 and Phase 2 of EXPO study 13 |
| Figure 2: Example 1 of Self-report and UDS results |
| Figure 3: Self-report and UDS example 1 outcome |
| Figure 4: Example 2 of Self-report and UDS results25 |
| Figure 5: Self-report and UDS example 2 outcome |
| Figure 6: Example 3 of Self-report and UDS results |
| Figure 7: Self-report and UDS example 3 outcome |

# 1. ACRONYMS AND DEFINITION OF TERMS

| Acronym | Meaning |
|-----------|-----------------------------------------------------------------|
| ADAPT | Addiction Dimensions for Assessment and Personalised Treatment |
| AD-SUS | Alcohol and Drug Service Use Schedule |
| AE . | Adverse Event |
| ALC-QFM | Alcohol – Quantity, Frequency and Maximum Consumption (ALC-QFM) |
| AR | Adverse Reaction |
| ARC | Addiction recovery clinic |
| BUP-SL | BUP-sublingual |
| BUP-SL-NX | BUP-Sublingual-Naloxone (Suboxone®) |
| BUP-XR | BUP- Extended-Release (US Sublocade®; prev. RBP-60000) |
| CEQ-F - C | Craving Experience Questionnaire (frequency version) (Cocaine) |
| CEQ-F — H | Craving Experience Questionnaire (frequency version) (Heroin) |
| CGI-I | Cfinical Global Impression (improvement) |
| CGI-S | Clinical Global Impression (severity) |
| CI | Chief Investigator |
| CONSORT | Consolidated Standards of Reporting Trials |
| CRA | Clinical Research Associate |
| CTIMP | Clinical Trial of Investigational Medicinal Product |
| СТИ | Clinical Trials Unit |
| CUD | Cocaine Use Disorder |
| DERS-SF | Difficulties in Emotion Regulation Scale – Short Form |

| DSM5 | Diagnostic and Statistical Manual of Mental Disorders 5th Edition |
|---|---|
| DMC | Data Monitoring Committee |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| ESP | ESPranor® |
| EQ-5D-5L | EurolQol Health Status (5 level) |
| EXPO | Extended-release Pharmacotherapy for Opioid Use Disorder |
| GCP | Good clinical practice |
| GLM | Generalised Linear Model |
| HEAP | Health Economics Analysis Plan |
| IMP | Investigational Medicinal Product |
| ITT | Intention to Treat |
| KCF | Keyworker Contact Form |
| LFT | Liver Function Tests (AST, ALT, albumin and bilirubin) |
| MET | METhadone (oral) |
| mITT | modified Intention to Treat |
| MoCA | Montreal Cognitive Assessment |
| NHS | National Health Service |
| NWORTH | North Wales Organisation for Randomised Trials in Health |
| OUD | Opioid Use Disorder |
| PRO-I | Patient Reported Outcome (improvement) |
| PRO-S | Patient Reported Outcome (severity) |
| PSI | Personalised Psychosocial Intervention |
| QIDS-SR | Quick Inventory of Depressive Symptomatology |
| SAE | Serious Adverse Event |
| SAP . | Statistical Analysis Plan |
| SAR | Serious Adverse Reaction |
| SCID-5-RV | Standard Clinical Interview for Dependence – Research Version (DSM-5) |
| SD | Standard Deviation |
| SURE | Substance Use Recovery Evaluator |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TLFB | Timeline Follow Back |
| TMG | Trial Management Group |
| ТОР | Treatment Outcomes Profile |
| TSC | Trial Steering Committee |
| UDS | Urine drug Screen |
| USA | United States of America |
| VAS-N (H/C) | Visual Analogue Craving Rating (Need) (heroine/cocaine) |
| VAS-W (H/C) | Visual Analogue Craving Rating (Want) (heroine/cocaine) |
| VIF | Variance Inflation factor |
| WSAS | Work and Social Adjustment Scale |

### 2. STATISTICAL ANALYSIS PLAN AUTHORSHIP

This SAP has been authored by Rachel Evans, Trial Statistician for the EXPO study, (Senior statistician NWORTH CTU) with input from CI, Mike Kelleher, Co-lead Investigator, John Marsden, Joanna Kelly and Caroline Murphy. Jatinder Bisla, EXPO Trial Manager and Zoë Hoare, Senior Trial Statistician for the trial (Principal Statistician NWORTH CTU).

Zoë Hoare (ZH Senior Trial Statistician) will remain blind throughout the conduct of the trial until the main analysis has been completed. Rachel Evans (RE) will be unblind for the purposes of reporting to the DMC. The draft plan has been circulated to the DMC members and TSC members for input and review prior to sign off.

### Statistician Blinding

Upon review of the protocol, it was noted that group numbers have been listed since protocol version 1.1. The Senior Statistician had reviewed and approved these protocols and the use of these group numbers could potentially unblind them to the treatment groups. These codes appear to be unblind with group 1 and 2 relating to phase 1 and groups 3 and 4 relating to phase 2.

It has not been confirmed either way which group these relate to explicitly however to ensure that the Senior Statistician remains blind to the data for analysis, the Trial Statistician will relabel the groups prior to analysis. The data using this relabelling will be used by the Senior Statistician to ensure blinding is maintained. All work will follow a full audit trail and documented in line with NWORTHs SOPs and MHRA guidance.

### 3. INTRODUCTION

### 3.1 BACKGROUND AND DESIGN

### **Background**

Daily doses of sublingual (tablet) buprenorphine hydrochloride (BUP-SL) and oral (liquid) METhadone hydrochloride (MET) are the first-line, standard-of-care (SOC) maintenance pharmacotherapies for OUD. MET is an opioid agonist with actions predominantly at the endogenous μ-opioid receptor. BUP is an opioid partial agonist/antagonist with actions predominantly at the endogenous μ-opioid and k (kappa) opioid receptors. In the UK, two other licensed BUP medications are also available for OUD — buprenorphine-naloxone (buprenorphine hydrochloride-naloxone dihydrate; Suboxone®; sublingual tablet; BUP-NX)

and buprenorphine-lyophilisate; ESPranor \*; sublingual wafer; ESP). BUP-NX contains the opioid antagonist naloxone (1:4 ratio with BUP) as a deterrent to injection of non-medical opioids. Indivior developed a subcutaneously injected, extended-release formulation of BUP (RBP6000). RBP6000 releases BUP for a minimum of 28 days, thereby facilitating monthly maintenance dosing. RBP6000 is now licensed as Sublocade\* in the USA (BUP-XR herein).

### Design

The EXPO study will determine the effectiveness of BUP-XR in a head-to-head superiority comparison with BUP-SL/MET (phase 1) and with an adjunctive psychosocial intervention (PSI) (phase 2) in the pragmatic context of specialist community setting addiction treatment programmes in England and Scotland provided by the NHS.

The Trial is a Phase III (CTIMP; IMP open-label, oral IMP comparators [no placebo]), multicentre, pragmatic, two-phase, randomised controlled trial. With a target total sample of 604 patients with Opioid Use Disorder (OUD; moderate-severe; DSM5), participants are allocated to one of four trial arms:

- BUP-XR
- BUP-SL/MET (including BUP-SL-NX and ESP)
- BUP-XR + PSI
- BUP-SL/MET (including BUP-SL-NX and ESP) + PSI

As BUP is the active component of BUP-SL-NX and ESP they will be categorised under BUP-SL within the remainder of this SAP and for analysis between trial arms.

### **Treatments**

BUP extended-release depot injection (USA Sublocade®; BUP-XR) is administered by subcutaneous injection into abdominal tissue. BUP-XR is available as a 100mg/0.5ml and 300mg/1.5ml pre-filled syringe. In EXPO, the drug is administered as two initial doses of 300mg given a minimum of 21 days apart, followed by 4 x 100 mg monthly maintenance doses.

Within the regimen and if the benefits are judged to outweigh the risks: (1) The 100 mg maintenance dose may be increased and maintained to 300mg if there is unsatisfactory clinical response (i.e. dose 3-6); (2) A 300 mg maintenance dose (i.e. dose 4 and 5) may be

reduced to 100 mg according to clinical assessment; (3) BUP-SL (including BUP-SL-NX and ESP) will be given on a rescue basis for patients who do not achieve a satisfactory clinical response to BUP-XR.

### Active comparator product(s);

- (1) BUP-SL (sublingual [tablet] BUP-SL), or substitute 4:1 ratio BUP-SL/naloxone 'Suboxone' [BUP-SL-NX]) usual dose 12-24mg/day; or substitute oral lyophilisate ESPranor (ESP) usual dose 9-18mg/day) are longstanding standard-of-care maintenance pharmacotherapy for OUD in the NHS;
- (2) MET (oral methadone hydrochloride; usual dose 60-120mg/d), longstanding standard-of-care maintenance pharmacotherapy for OUD in the NHS.

### Trial Phases

The study consists of two phases. Phase 1 of the study refers to the analysis of BUP-XR and BUP-SL/MET and phase 2 refers to the analysis of BUP-XR + PSI and BUP-SL/MET + PSI. There will be separate statistical analysis plans for the two study phases. Recruitment in phase 1 of the study is on a 1:1 allocation ratio to BUP-XR and BUP-SL/MET across 4 clinical recruitment sites in the West Midlands, Greater Manchester, Newcastle and Tayside. During phase 1, the South London site will recruit to groups on a 4:4:1:1 allocation ratio for approximately 6 months whilst resources are in place to allow more participants to be allocated to psychosocial therapy (e.g. therapists in post). During the subsequent approximate 18 months of recruitment, there will be a 1:1 allocation ratio to BUP-XR + PSI and MET/BUP-SL + PSI (only at the South London site). The timescales for these ratios may change depending on recruitment levels and resource availability. Figure 1 below represents the study's randomisation structure across sites. The current statistical analysis plan (SAP) only concerns phase 1 of the study.



Figure 1: Randomisation summary for Phase 1 and Phase 2 of EXPO study

### **Analysis set**

Primary analysis will be conducted on an intention to treat (ITT) basis, defined as all participants that are randomised are analysed as allocated, regardless of their treatment.

Certain circumstances may occur that result in randomised participants not being analysed. Such circumstances can arise if patients are randomised in error, e.g.

- If the same participant is mistakenly randomised twice
- If an ineligible patient is randomised and must be withdrawn from the study Eligibility
   violations

If any post randomisation eligibility violations are identified, the study team along with the sponsor and independent committees will establish whether the participant can remain in the study. For cases where the criteria violated does not affect clinical outcome or patient safety these participants will be kept in the ITT analysis set. Sensitivity analysis will be conducted

removing eligibility violations by conducting a modified intention to treat (mITT) analysis, see section 6.9 for more details.

All exclusions due to randomisation errors or eligibility violations will be reported clearly.

### **3.2 TRIAL OBJECTIVES**

### **Primary Objective:**

During six months of active trial treatment, the primary objective of this superiority study is to determine the difference in effectiveness (in terms of reduced use of heroin and illicit opioids) of BUP-XR and either MET or BUP-SL. Study participation will be offered to patients already enrolled in BUP-SL and MET maintenance treatment.

With a 1-week measurement grace period from randomisation, the primary endpoint is the count of days abstinent from heroin and illicit opioids during six months of treatment combined with urine drug screen samples which are negative for non-medical opioids.

## **Secondary Objectives:**

To explore study group differences on the following measures:

- \*Clinical superiority of BUP-XR plus PSI versus BUP-SL/MET plus PSI;
- (2) Safety of BUP-XR;
- (3) Treatment retention;
- (4) OUD and CUD remission status;
- (5) Clinician rated impression of patient response to treatment;
- (6) Patient reported recovery outcomes;
- (7) Mediation of craving, depression, work and social adjustment, and cognitive function on outcome.

\* Secondary Objective (1) not covered by this SAP as is part of phase 2 analysis.

Additionally, longer-term outcomes will be collected through data-registry indicators of criminal convictions and health service utilisation. The analysis of these outcomes are not included in this SAP.

### 3.3 CONSORT DIAGRAM

# **CONSORT 2010 Flow Diagram**



4. STATISTICAL PRINCIPLES

4.1 SAMPLE SIZE JUSTIFICATION

The required number of participants has been estimated using that required for a Poisson

regression model taking a baseline rate of 0.6 (60% abstinent days per month) and assuming

a 23% target difference in the count of days of abstinence from heroin over the study period

of 161 days. This target difference is informed by results of the ARC trial (ISRCTN69313751):

56.78% for the treatment-as-usual control (i.e. assuming 17 abstinent days over a period of

28 days).

To obtain 90% power, for a Poisson regression, with alpha at 5% and with 15% inflation for

attrition, EXPO has a target total of 304 participants for the statistical comparison of the

primary outcome recorded for BUP-XR and MET/BUP-SL.

A sensitivity check on the power calculation on the assumption of a greater response has been

completed. With a sample of 304 subjects and a 23% target difference achieved, a higher

baseline rate of 0.75 observed would achieve 97.5% statistical power.

Additionally, a sensitivity check has been conducted assuming a reduced baseline rate. With

a sample of 304 subjects and a 23% target difference achieved, a baseline rate of 0.5 observed

would achieve 88% statistical power.

A power analysis will be completed as part of the main analysis for the study.

4.2 RANDOMISATION

Online randomisation system will be provided by King's CTU. Randomisation procedure will

be on a 1:1 allocation ratio by stratified block with random varying block sizes, stratified for

Centre (West Midlands, Manchester, Newcastle and Tayside) and Current (last 28 days) drug

injecting status (yes/no). At South London for approximately the first 6 months (subject to

change depending on resource and recruitment rates) of recruitment, patients will be

randomised to one of four groups on a 4:4:1:1 allocation ratio, with Current (last 28 days) drug

injecting status (yes/no). Figure 1 in section 3.1 portrays this.

Statistical Analysis Plan for EXPO Phase 1 Version 4 Date 08/06/2022 Page | 16

Justification for these stratification factors is as follows: (a) site is required for the random-effects model; (b) it is expected that there will be relatively poorer outcome among participants who are drug injectors. The randomisation procedure will use stratified random blocks of varying size to ensure even allocation.

### 4.3 LEVELS OF CONFIDENCE AND P-VALUES

All statistical tests for the primary endpoints will be two-sided and will be performed using a 5% significance level. Confidence intervals for estimated effects will be presented as 95% and two-sided.

Secondary outcomes will not be adjusted for multiple comparisons, as standard. The primary outcome is powered for at the significance level stated. Analysis of all secondary outcomes is considered exploratory, and any statements of results related to these outcomes will be reported appropriately. 95% confidence intervals will be reported along with the p-value of the effect.

### **4.4 ADHERENCE**

BUP-SL (including BUP-SL-NX and ESP) (active sublingual comparator): The usual dose is 12-24mg/day (ESP usual dose 8-18mg/day). Clinical practice in NHS clinics is supervised (directly observed dosing) in a community pharmacy followed by provision of patient self-administered 'take home' doses according to clinical response (i.e. informed by negative urine drug screens [UDS]; adherence to prescription; retention in treatment).

**MET** (active oral comparator): The usual dose is 60-120mg/day. Clinical practice in NHS clinics is supervised (directly observed dosing) in a community pharmacy followed by provision of patient self-administered 'take home' doses according to clinical response (i.e. informed by negative UDS; adherence to prescription; retention in treatment).

Adherence to the intervention will be reported descriptively using the BUP-XR Injection Log and for the comparator the BUP-SL/MET Medication Record form and UDS. This will include injection frequencies, patterns of dosage (i.e. injection size in mg), oral medication frequencies and patterns of dosages.

### 4.5 PROTOCOL VIOLATIONS

Definition of protocol violations and deviations. Violation is an intended failure to adhere to the protocol such as wrong treatment being prescribed or administered or incorrect data being collected and documented. A protocol deviation is an unintended failure to adhere to the protocol and examples include errors in applying inclusion/exclusion criteria or missed follow-up visits due to error. Per protocol analysis is not planned for the study but deviations and violations will be monitored and reported throughout the study and detailed descriptively in the analysis report. If protocol deviation occurrences rise above 10% then sensitivity analysis as detailed in section 6.5 will be conducted. Some examples of protocol deviations which might occur in this study include;

- Patients not receiving randomised allocation
- Patients not receiving treatment within 7 days
- Ineligible participants being randomised

### 4.6 MISSING DATA

Primary and secondary count-based measures For the count-based measures two situations of missing are expected. Firstly, there will be those who have missing observations periodically through the study observation period but have remained in the study for these patients multiple imputation as described above will be adopted. The memory recall for the TLFB is 3 months therefore if a patient hasn't been to visits for a couple of months recall of up to 3 months is deemed reliable [4 - 6]. Where patients have gaps in their recall on the primary outcome (at most this would be 3 months) we would use the available data to impute for the patient. Sensitivity analysis will be conducted on this imputation using a best-case worst-case analysis, see section 6.9 for more details.

Secondly, there will be some cases of participants who completely drop out of the study during the observation period i.e. withdrawals or loss to follow ups. For these patients on the primary outcome and secondary count-based measures an offset (censoring) will be used to represent different exposures rather than multiple imputation.

Furthermore, some of the primary and secondary end points (TLFB) are based on self-report and UDS tests. Where data is available for self-report and UDS, if the results are inconsistent the UDS data will override the self-report, as indicated in section 5.2. Essentially where UDS is not available this does not result directly in missing data for the outcome as the self-report

will provide this data. However, the reliability of the self-report may be impacted therefore sensitivity analysis on missing UDS data will be conducted, see section 6.9 for more detail.

### Continuous outcome measures

Missing observations are expected within the dataset. For missing items within an outcome measure, the published rules for completing missing data for the relevant measure will be applied. Where there are no missing data rules for the measure, if the number of missing items on an outcome is 20% or less, then the missing value for the item will be substituted by the individual's mean score for the remaining items on the scale (Bono, Ried, Kimberlin and Vogel 2007). If there are more than 20% missing items in the scale the outcome measure will not be calculated for the participant at that time point and multiple imputation methods will be used.

Predictive mean matching multiple imputation methods will be adopted for an outcome measure total score if missing data arises above 5%. For multiple imputations, the number of imputations completed will be dependent upon the percentage of missing data [2]. The missing outcome measures will be imputed using group allocation and stratification variables along with any baseline characteristics that are deemed to be predictors of missingness. Baseline characteristics will be assessed for being predictors of missingness by running statistical tests on completers versus non completers and evaluating if any differences are present between the two.

Baseline factors to be assessed as predictors of missingness include;

- Centre
- Current injecting status
- Length of current treatment episode
- Preference of MET or BUP-SL
- Use of cocaine in the past month
- Sex at birth
- Age
- \*Ethnicity
- Baseline outcome scores on the following measures:
  - o QIDS-SR
  - WSAS
  - PRO-S

o ALC-QFM

ADAPT (all subscales)

\*Ethnicity is being collected with five categories - Black, White, Mixed, Asian and other. Depending on the prevalence of responses in each of these categories, the variable will be treated either with all 5 categories as collected or if appropriate will be dichotomised into 'White' and 'Non-White' if the range across categories are low.

### 4.7 ASSUMPTION CHECKING

All assumptions relating to the models will be checked and evaluated whether appropriate to use with the data. If any of the assumptions are substantially violated then appropriate non-parametric tests will be conducted. Appendix 4 contains details of the assumptions associated with each model and the methods to be used to assess these assumptions.

Outliers or unusual values will be assessed by running Grubbs [7] test for outliers and visually inspecting a boxplot. No outliers will be discarded if they are within plausible range. Primary analysis will be conducted keeping the outliers in the dataset and if necessary, sensitivity analysis will be conducted by removing the outliers and evaluating any effects on the results and conclusions of analysis. Any outliers removed will be fully reported.

The distribution of the data will be checked. For the count data a decision will need to be made as to which analysis method to use for the outcome based on the distribution of the data. Appendix 1 contains a flow diagram to be followed to decide which analysis model is to be run based on the data distribution.

For continuous data a decision will be made as to whether a transformation should be applied to the data and if so which transformation should be used. If transformation is required the distribution of the transformed data will be checked. Analysis will be reported on the original scale, transforming variables back. If a transformation is inappropriate then non parametric analysis methods will be considered.

For the logistic regressions, if detection rates (number of responses observed) are very low, where appropriate, either a Firth's Bias-Reduced Logistic Regression will be conducted or descriptive statistics reported.

5. DATA

KCTU MACRO database;

All baseline and follow-up data will be entered on the online InferMed MACRO electronic data

capture (EDC) system (infermed.com). This system is regulatory compliant (GCP, and the EC

Clinical Trial Directive). An electronic case report form (eCRF) using the MACRO EDC will be

programmed by the KCTU and hosted on a dedicated secure server. The eCRF system will have

full audit trail, data discrepancy functionality, database lock functionality, and supports real

time data cleaning and reporting. The Trial Manager will request usernames and passwords

to any new researchers. Only those authorised by the Trial Manager will be able to use the

system.

After written recording, each research worker will aim to transcribe data onto the eCRF within

one working week of a participant assessment. After completion of all follow-ups and prompt

entry of data, the Clinical Research Associate (CRA) will review the data and resolve queries

with sites. At the end of the trial, each centre will be supplied with their eCRF data for storage.

This will be filed locally for any future regulatory or internal audit.

Database lock for phase I will be undertaken within approximately 3 months of last patient,

last visit and will be controlled by TMG of participants enrolled in groups 1 and 2. Database

lock for phase II will be within approximately 3 months of last patient, last visit and will be

controlled by TMG of participants enrolled in groups 3 and 4. This will be once the data has

been monitored, all queries resolved and PI sign off has been obtained for participants in the

BUP-XR and BUP-SL/MET (including BUP-SL-NX and ESP) arms.

KCTU Randomisation System;

The King's Clinical Trials Unit Randomisation system will be used in EXPO. This will be a secure

password-protected, web-accessed system.

Once a patient has consented and it is confirmed that all potential medication is in place within

the next 7 days, all baseline data collected and eligibility confirmed, the staff member will log

Statistical Analysis Plan for EXPO Phase 1 Version 4 Date 08/06/2022 Page | 21

into the randomisation system (www.ctu.co.uk) and randomise the participant, detailing the relevant stratification factor information;

- \*(a) Site (South London, the West Midlands, Greater Manchester, Newcastle and Tayside)
- (b) Current (last 28 days) drug injecting status (yes/no)

\*Note there are four systems built for the study three for South London and one for the other sites.

1 system for other sites at 1:1 ratio XR BUP-SL and MET/BUP-SL

1 system South London at ratio 4:4:1:1 BUP-XR, MET/BUP-SL, BUP-XR + PSI, MET/BUP-SL + PSI

1 system South London at ratio 1:1:1:1 BUP-XR MET/BUP-SL, BUP-XR + PSI, MET/BUP-SL + PSI

1 system South London at ratio 1:1: BUP-XR + PSI, MET/BUP-SL + PSI

The randomisation procedure will use stratified random blocks of varying size to ensure even allocation. See section 4.2 for more details on randomisation.

### **5.1 TIME POINTS OF OUTCOMES MEASURES**

Table 2 indicates the data and study measures to be collected during the trial and at which time points across the study they are collected.

Table 1: List of outcome measures to be collected and time point of collection

| Measure | Baseline | Randomisation | Ongoing | Week 1 | Week 2 | Week 4 | Week 6 | Week 8 | Week 10 | Week 12 | Week 14 | Week 16 | Week 18 | Week 20 | Week 22 | Week 24 | Withdrawal | Week 24<br>onwards | Ext. Phase<br>Interview +++ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Consent § | Х | | 222 | | | | | | | | | | | | | | | Х | X |
| | X | Н | | _ | | | | | | | $\vdash$ | - | - 6 | | | | | - | |
| Screening<br>UDS | ^ | Н | | _ | Х | Х | Х | X | Х | Х | Х | Х | Х | Х | Χ | Х | X | | |
| | | | | 7. | ^ | | ^ | ^ | | | ^ | _ | | | ^ | | ^ | 4.866 | E 1/2" |
| LFT * | Х | Ш | | 2 | | Χ | | | | Χ | | | | | 7 | Χ | AT S | X | |
| BUP-XR** | | | | Х | | Χ | | X | | Χ | | Χ | | Χ | 134 | | 200 | Х | |
| BUP-SL/MET ** | | 9 | X | | | | | | | 4 | | | | | | | White | 1920 | |
| ALC-QFM (TOP)*** | X | | | = | | | | - | | | | | | | Ш | Χ | 3.0 | | - |
| SCID-5-RV | Х | | | | (0) | | | | - | X | | | | | | X | | 18-51 | X |
| ADAPT | X | | | | | Х | | | | Χ | | | | | | Х | 1000 | | 4 |
| CGI-S | X | | | | | - | s | | | 22 | | | 0 | 2 | | | 226. | SEN | 4.00 |
| CGI-I | | | | | | Х | | | 8 | X | | | | | | Χ | | 250 | |
| CEQ-F H*** | X | | | | - | Х | | Х | | Х | P | Χ | 10 | X | | X | X | TOTAL | |
| CEQ-F - C*** | Х | | | 22 | | Χ | | Х | | Χ | 0 | Х | | Χ | | Χ | X | DATE | |
| VAS-N (H/C)*** | Х | | | 50 | 0 | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | X | 1715 | Best |
| VAS-W (H/C)*** | Х | | | | | Х | | Х | | Χ | | Χ | | Х | | Χ | X | 17.60 | 2220 |
| DERS-SF | Х | | | | | Χ | | | | Χ | | | | | | X<br>X<br>X<br>X<br>X<br>X | | | X |
| WSAS | Х | | 8.5 | | | Х | | | | Χ | | | | | | Χ | | E:-0X | |
| EQ-5D-5L | Х | | | n | | | | | | X | | | | | | Χ | | | Party. |
| AD-SUS | X | 5 | | | | | 54 | n e | | Х | | | | | | X. | | | |
| KCF*** | | 90 | | | | Х | | 11 | | Х | | | | | | Χ | | 2 14 50 | |
| QIDS-SR | X | | 2/2 | | 0 | Х | | | | Χ | | | | | | Χ | | 25/62 | |
| SURE | | | | | | Х | | | | Х | | | | | | Х | | -512.6 | |
| PRO-S | X | | | | | | | | | | | | | | | | MER | FERE | |
| PRO-I | | | | | | Х | | | | Х | | | W | | | Χ | Tekto | 14200 | 400 |
| MoCA*** | X | | 015 | | | | | | | Х | | | | | | | <b>3</b> 77.07 | Ref 34 | 5.73 |
| OSTQOL | | | | | | | | | | | | | | | | | BH IS | 262 | X |
| PHQ-4 | | | 70 | | | | | | | | | - 1 | | | | | 9.4 | 215.20 | X |
| PHQ-15 | | | 1 | 2 | | | | | | | | 10 | | | | | | E-012 | X |
| Exit Interview+ | | | Ve. | | 7/ | | | | | | | | | | | Χ | 527 | 4"57 | |
| BUP-SL/MET + PSI | | | | 2 , | | | | | | | | | | | | X | 500 | | |
| Interview++ | | | 338 | | | | | | | 36 | | | | | | | 2-10 | | |
| TLFB | X | | X | 3 /3 | ii . | | | | . 25 | | | (6) | | | | 5 | | 65 S. | X |
| Con Meds**** | | Γ | X | | | Х | | | | Х | | | | | | Χ | | X | |
| Adverse Events Log | 1 12 | | X | | | | | | | | | | | | | | 1 | X | 1042 |
| Research Payments | Х | | | Х | Х | X | Х | Х | Х | Χ | Х | X | X | Х | Х | X | | THE REAL PROPERTY. | X |
| **** | 20 | | | 10 | 10 | 10 | 5 | 10 | 1 0 | 10 | 5 | 10 | 10 | 10 | 5 | 10 | | | 20 |

§ screening to include pregnancy test, demographics and medical history. Participants receiving XR- BUP-SL reconsented once at week 24 to continue receiving monthly injections;

\* LFT for all participants at screening; during treatment for BUP-XR participants only under protocol;

<sup>\*\*</sup> refer to section 6 of the protocol for guidelines;

\*\*\* used for mediation model;

\*\*\*\* ConMeds to be recorded continuously and reviewed at week 4, 12 and 24;

<sup>\*\*\*\*\*</sup> research payments are time offset to attend the clinic to complete research measures and cover travel (either a £20, £10, or £5 value, as detailed per visit applicable; loaded onto a prepaid card).

<sup>+</sup> Exit Interview conducted at South London, Newcastle, West Midlands and Tayside sites with BUP-XR participants only. Participants will be reimbursed an additional £20 for their time in taking part in the interview (loaded onto a prepaid card).

<sup>++</sup> BUP-SL/MET +PSI Interview conducted at South London with BUP-SL/MET +PSI participants only. Participants will be reimbursed an additional £20 for their time in taking part in the interview (loaded onto a prepaid card).

<sup>+++</sup> Extension Interview conducted at the South London and Newcastle sites with BUP-XR participants who consented to continue treatment after week 24 between 12-24 months of them being randomised in the trial.

### 5.2 DEFINITIONS AND CALCULATIONS OF OUTCOME MEASURES

The following outcomes measures have been identified in relation to the objectives as described in section 3.2

### Primary objective;

### Objective 1 - effectiveness of BUP-XR and MET/BUP-SL

Measure 1; Number of days abstinent from 'substance' during days 8-168 (weeks 2 to 24, 161 days); combining self-report information from time-line follow-back interview adapted from the Treatment Outcomes Profile and incorporating data from 12 scheduled urine drug screens (UDS). The UDS results will provide biological verification for up to 36 out of the 161 days required.

- Days abstinent from illicit/non-medical opioids (Primary outcome)
- o Days abstinent from cocaine (secondary outcome)
- o Days abstinent from benzodiazepines (secondary outcome)

The primary outcome will be determined by combining the self-report results and UDS results to give an overall count for each participant. Where data is available for self-report and UDS, if the results are inconsistent the UDS data will override the self-report. Where this occurs, the result will overrule the self-report for the day of the UDS and the two days prior. Examples are indicated below.

### Example 1

A negative self-report for 4 days, day 4 a positive UDS, figure 2 below.

| | Day 1 | day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | Day 10 |
|---|---|---|---|---|---|---|---|---|---|---|
| Self-report | no drug use | no drug use | no drug use | no drug use | drug use | drug use | drug use | drug use | drug use | drug use |
| UDS (Day 4) | | W II | | positive | | | | | | |

Figure 2: Example 1 of Self-report and UDS results

The UDS would trump the 'no drug use' self-report for days 2-4, resulting the outcome in figure 3.

| | | Day 1 | day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | Day 10 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Outco | me: | no drug use | drug use | drug use | drug use | drug use | drug use | drug use | drug use | drug use | drug use |

Figure 3: Self-report and UDS example 1 outcome

### Example 2

A positive self-report for 2 days, day 4 a negative UDS as shown in figure 4.

| | Day 1 | day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | Day 10 |
|---|---|---|---|---|---|---|---|---|---|---|
| Self-report | no drug use | no drug use | drug use | drug use | drug use | drug use | drug use | drug use | drug use | drug use |
| UDS (Day 4) | | | | negative | | | | | | |

Figure 4: Example 2 of Self-report and UDS results

The negative UDS would trump the self-report for days 2-4 (day 2 no change) resulting in the outcome below in figure 5.

| 0 | Day 1 | day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | Day 10 |
|---|---|---|---|---|---|---|---|---|---|---|
| Outcome: | no drug use | no drug use | no drug use | no drug use | drug use | drug use | drug use | | drug use | drug use |

Figure 5: Self-report and UDS example 2 outcome

### Example 3

UDS and self-report align figure 6, therefore no change to the outcome in figure 7

| | Day 1 | day 2 | Day 3 | Day 4 | Day 13 | Day 14 | Day 15 | Day 16 | Day 17 |
|---|---|---|---|---|---|---|---|---|---|
| Self-report | drug use | drug use | drug use | drug use | no drug use | no drug use | no drug use | no drug use | drug use |
| UDS (Day 4 and day 16) | 7 | | = | positive | 97 | | | negative | |

Figure 6: Example 3 of Self-report and UDS results

| Outron | | Day 1 | day 2 | Day 3 | Day 4 | Day 13 | Day 14 | Day 15 | Day 16 | Day 17 |
|---|---|---|---|---|---|---|---|---|---|---|
| Outcom | 3; | drug use | drug use | drug use | drug use | no drug use | no drug use | no drug use | no drug use | drug use |

Figure 7: Self-report and UDS example 3 outcome

The syntax for calculating this variable will be validated and verified fully prior to database lock.

During a data review it was identified that some participants had been called in for their last visit early, resulting in the full primary outcome of 161 days not being obtained. The participants in question are not lost to follow up or withdrawals and are just missing due to an administration error and in most cases only by a day or two. It was noted that patient records could provide data for some of these missing days therefore, with input from independent committees, it was decided that for the TLFB data some of the final follow up days are being input based on these medical notes.

Where the TLFB data is not obtainable from the patient notes, the missing days will be imputed using a devised rule. The missing data rule used for these missing days will look at the last 14 days of data that are available for the participant, the percentage of drug use will be calculated. For all missing days a random number will be generated (either a 0 or 1, no use or use) using a probability based on their percentage used in the last 14 days.

Measure 2; Longest time in days *continuously* abstinent from 'substance' during days 8-168 (weeks 2 to 24, 161 days); combining self-report information from time-line follow-back and 12 urine drug screen (UDS) results.

- Longest count of days continuously abstinent from illicit/non-medical opioids
- o Longest count of days continuously abstinent from cocaine
- Longest count of days continuously abstinent from benzodiazepines

### Secondary objectives;

Objective 1 – Clinical superiority of BUP-XR plus PSI versus BUP-SL/MET plus PSI.

Will be analysed as part of phase 2 of the study and detailed in a separate SAP

### Objective 2 - Safety profile

Tabulation of AEs, ARs, SAEs, SARs and SUSARs in each group

# Objective 3 - Treatment retention

- Measure 1; Total retention time Days enrolled in maintenance medication for opioid use disorder (OUD) from first day following grace period (day 8) to day 168 (across 161 days weeks 2 to 24)
- Measure 2; Survival time Days from randomisation to first discontinuation (i.e. time (days) enrolled in study treatment).
- \*Measure 3; Time (days) enrolled in study treatment (retention) from week 24 to date last participant randomised plus 9 months.

\*Measure 3 Will be analysed as part of the extended phase of the study and detailed in a separate SAP

# Objective 4 OUD and CUD remission status

- Assessed by Standard Clinical interview for Dependence research version (SCID-RV)
  - o Remission status (Yes/No) at 12 weeks
  - o Remission status (Yes/No) at 24 weeks

# Objective 5 Clinician rated impression of patient response to treatment (at 24 weeks)

- Measure 1; Clinical Global Impression scale (severity and improvement CQI-S/CGI-I)
- Measure 2; Addiction Dimensions for Assessment and Personalised Treatment (ADAPT)

### Objective 6 Patient reported recovery outcomes (at 24 weeks)

Measure 1; Craving response using Craving experience questionnaire (CEQ-F)

Measure 2; Visual analogue craving rating (Need) (VAS-N)

Measure 3; Visual analogue craving rating (Want) (VAS-W)

Measure 4; Social functioning using Work and Social Adjustment Scale (WSAS)

Measure 5; Depression using Quick inventory of Depressive Symptomatology (QIDS-SR)

Measure 6; Improvement and Recovery using Substance Use Recovery Elevator (SURE)

Measure 7; Patient Reported Outcome Status (severity and improvement - PRO-S/PRO-I)

Measure 8; Emotion regulation using Difficulties in Emotion Regulation Scale short form (DERS-SF)

**Measure 9;** Alcohol quantity, frequency, maximum consumption (ALC-QFM (TOP) - quantity and frequency only - maximum will be reported descriptively).

### **Objective 7 Mediation analysis**

Mediation of craving, work and social adjustment, and cognitive function on outcome.

### Mediator measures;

- Visual analogue scale (VAS) for the perceived need and want for non-medical opioids and cocaine (VAS-N and VAS-W)
- Craving Experience questionnaire, frequency version (Heroin) (CEQ-F-H)
- Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR)
- Montreal Cognitive Assessment (MoCA)
- Work and Social Adjustment Scale (WSAS)

### Moderator measures;

Sex at birth

- Age
- Current injecting status
- Centre
- Measure/Outcome baseline

Separate models will be run for each of the mediator measures using the moderator measures listed above, therefore, in total five models will be evaluated (i.e. baseline and each mediator)

### **Other Measures**

Appendix 2 contains further details of each outcome measure and Appendix 3 contains scoring details for the relevant measures.

Many of the measures are being collected across several time points during the study, as indicated in table 2 but are only being primarily analysed here at 24 weeks. Exploratory analysis of the secondary outcomes collected at all time points other than the primary endpoint of 6 months will be detailed in a separate SAP. Additionally, the EQ5D-5L, AD-SU, PHQ-15, PHQ-4, OSTQOL and keyworker contact form are being collected but not analysed here. These measures will be used for health economic analysis and qualitative evaluation at a later date. Details on this analysis is to be included in a separate health economics analysis plan (HEAP) that will align with this SAP and signed off prior to data lock.

### **5.3 SAFETY DATA**

All adverse events, reactions and serious and unexpected events/reactions will be reported immediately following the procedure noted in the protocol (section 11.2). Safety data in the form of all AEs will be presented to the DMC on a scheduled basis. This report will cover the number of events and number of subjects affected split by treatment arm and categorised by seriousness (not serious, death, is life-threatening, requires hospitalisation or prolongation of hospitalisation, persistent or significant disability or incapacity, consists of a congenital anomaly or birth deficit, important medical event or pregnancy). Frequencies of system organ class will also be presented split by treatment arm. No statistical testing of these data will be undertaken in the DMC report. These data will also be included in the final analysis report. Precipitated withdrawal symptoms will be included in the discussion section of the primary paper as a narrative in relation to the Adverse Events table. This will not be a formal analysis but to check if there is a correlation between the first 24-48 hours prior to treatment and first

month after treatment and numbers of precipitated withdrawal symptoms reported between the treatment arms.

### **6. STATISTICAL ANALYSES**

### **6.1 ANALYSIS TIME FRAME**

Table 2: Planned target timeline for analysis dependent on recruitment period

| Task | *Updated following COVID recruitment pause |
|------------------------|--------------------------------------------|
| Last patient recruited | ~October 2021 |
| Final patient visit | ~May 2022 |
| Database Lock | ~June/July 2022 |
| Final Analysis | ~August 2022 |

<sup>\*</sup>The analysis timelines are dependent on recruitment rates, COVID-19 impacts and discussions with the funder. Delivery of the analysis report will require at least one month following database lock to complete.

### **6.2 BASELINE ANALYSIS**

Characteristics collected at baseline will be presented descriptively both overall and by treatment arm. No statistical testing of baseline differences will be completed, only used to assess balance. Categorical variables presented using counts and percentages, continuous variables with mean, SD and range.

### **6.3 INTERIM ANALYSIS**

There are no planned interim analyses and as such the study is not powered to achieve these. There are no planned stopping criteria based on efficacy and stopping based on safety will be guided by the DMC.

### **6.4 CONSORT ANALYSIS**

The patient flow information, as shown in section 3.4 above as advised by CONSORT reporting standards, will be completed with values relating to participants numbers. Additionally, data will be presented on screening, eligibility, recruitment, treatment discontinuation and withdrawn/lost to follow up presented for the entire study and split by recruitment site.

Where possible reasons for ineligibility or non-recruitment will be reported. From these data related eligibility, recruitment and retention rates will be calculated and presented in the final analysis report.

### **6.5 DESCRIPTIVE STATISTICS**

Descriptive statistics of the data will be presented in the final analysis report. This will include randomisation figures, demographics, other data characteristics of the outcome measures and data completeness levels. All will be presented overall and split by allocation group.

Figures will be presented for the Randomisation data by each stratification variable;

- Allocation group
- Centre
- Current injecting status

The following demographics and data characteristics will be presented;

- Sex at birth
- Age
- Ethnicity
- Preference of MET or BUP-SL
- Use of cocaine in the past month
- Length of treatment episode (in days)
- Age started opioid substitution therapy
- OUD medication length this episode
- Rescue medications required
- ALC-QFM (TOP) maximum consumption

Descriptive statistics of the outcome measures will be produced for the primary and secondary variables as listed in Appendix 2.

For all statistics, continuous variables will be reported with mean values, standard deviations and ranges. Categorical variables will be presented with counts and percentages. If data are not normally distributed then medians and interquartile ranges will be reported.

Graphical representations of the objective one measures (days abstinent and longest days) will be displayed to evaluate and observe where across the study patients 'relapsed/started using again' and where withdrawals in the study were common.

In addition, we will plot a cumulative distribution function for each group on the primary outcome, other graphical representations may be used for treatment effect visualisation.

### **6.6 ANALYSIS OF PRIMARY OUTCOME**

The primary outcome will be analysed using a Poisson regression model (i.e. generalized linear model with a log link) to assess the differences between the two treatment groups (BUP-XR or MET/BUP-SL). The randomisation stratification variables (centre and current injecting status) will be included in the model as covariates. If a Poisson distribution is not observed then the regression model to be used will be dependent on the distribution of the data and decided following the decision tree in appendix 1, figure 1.

### **6.7 ANALYSIS OF SECONDARY OUTCOMES**

All secondary outcomes are to be analysed as the primary outcome including the randomisation stratification variables (centre and current injecting status) in the models. The model used will be based on the outcome measure (dependent variable) format and the distribution of the data.

- Count variables will be analysed using a Poisson regression model. As with the
  primary outcome measure the exact model to be used will be based on the
  distribution of the data following the decision tree in appendix 1, figure 1.
- Continuous measures will be analysed with a GLM to assess the differences between
  the means of the treatment groups. In addition to the randomisation stratification
  factors, the baseline measure scores of the associated outcome will be included in the
  models as covariates to account for the baseline scores.
- · Binary variables will be analysed using a (binary) logistic regression model
- Ordinal variables will be analysed using an ordinal logistic regression model

Appendix 2 details the outcome measures to be analysed and their associated models.

A causal mediation analysis (including craving, MoCa, QUIDS-SR and WSAS as mediators in separate models) will be implemented using a counterfactual framework to include a treatment/mediator interaction and covariates, based on univariable path screening, and with bias corrected bootstrapped estimates.

### **6.8 SUBGROUP ANALYSES**

Subgroup analyses will be conducted for the primary objective/outcome on the following:

- Using cocaine (Yes/No)
- Length of time in treatment (less than one month/one month or longer)
- Benzodiazepine use past month to admission (Yes/No)
- CGI-S (Mild/Severe)

### 6.9 SENSITIVITY ANALYSES OR MODEL TESTING

Sensitivity analysis will be conducted on the primary analysis model including the variables that were identified as predictors of missingness as covariates in the model.

Additionally, sensitivity analysis may be required around any assumptions made for the primary analysis (e.g. outliers, data distributions) but will only be conducted if necessary. This will include a best-case worst-case analysis on the self-report missing data on the primary outcome. Best case would assume that patients did not use during any missing time periods and worst case would assume that they did use substances to evaluate any impact the imputed data may have had on the results.

Furthermore, the confidence of the reliability of the self-report will be checked by conducting a best-case worst-case sensitivity analysis on the UDS missing data for the TLFB outcomes. For those who have a missing UDS, we will assume all missing as negative for one dataset and then for another dataset assume all missing as positive. Utilising this best—worst case scenario will provide a range of values between which the real outcome is likely to lie. The width of this range is likely to be influenced by many factors (including the COVID pandemic and not being able to collect the UDS).

Primary and secondary analysis will be conducted on an ITT basis (including all those randomised to be analysed. Sensitivity analysis may be conducted, if necessary, on protocol deviations or eligibility violations by removing them from the analysis set. This includes protocol deviations (but is not limited to) such as;

Patients not receiving randomized allocation (per protocol analysis)

Patients not receiving treatment within 7 days (per protocol analysis)

Ineligible patients being randomised (mITT analysis)

Sensitivity analysis will be conducted on the patient's months in treatment (for current

episode) at baseline by running the model including the variable as a factor.

Additionally, sensitivity analysis of the patient's preference of BUP-SL or MET will be

conducted again by running the model including that variable as a factor. This will be

conducted given that there is an adequate sample of data per group at each level of the

variable (BUP-SL or MET) a sample of 50% - 60% in the MET group will indicate that we will

run this sensitivity analysis.

Sensitivity analysis will be conducted truncating at 14 days at the end of the TLFB data (i.e.

day 8 - day 154) to assess the impacts of using the medical notes due to the administration

error highlighted in section 5.2.

Furthermore, there will be a sensitivity analysis around the week 'Grace period' of the primary

outcome where we will include all TLB data from day 0 to day 168.

COVID-19

A sensitivity analysis around the impact of the COVID-19 pandemic has been considered. The

biggest impact the pandemic has had on the trial, to date, is the pause in recruitment which

occurred March 2020 to July 2020, however, the trial is currently back recruiting in all sites.

Some of the psychosocial intervention was delivered remotely (by telephone and video call)

and some data collection was collected remotely during this time. The paper will include a

summary of milestone dates such as the date COVID-19 was declared a pandemic by the World

Health Organisation, date the Government imposed lockdown and dates the trial paused and

restarted recruitment.

In addition, during the pandemic, changes to the distribution of medication for those in the

oral arms of the study occurred. National clinical guidance was issued on 22 May 2020

Statistical Analysis Plan for EXPO Phase 1 Version 4 Date 08/06/2022 Page | 33

indicating that rather than daily medication collection participants were to collect weekly and not be observed whilst taking them. This may have had an impact on some participants as they had access to more medication and more freedom with these (i.e. there was be choice as to whether to take medication as directed). This could result in participants in these groups being more likely to disengage from treatment and relapse. However, subsequent guidance has recommended that supervision and dispensing interval should return to be determined on a case-by-case basis and informed by risk assessment [8]. This advice may change again in the event of a substantial increase in Covid-19 infection incidence.

Although these changes may have had an impact, investigators have no reason to believe that this will affect any signal (or no signal) detected.

However, baseline characteristics will be summarised by enrolment period (pre Covid-19, during Covid-19, post Covid-19) to assess if there are any relevant differences in the recruited population relative to the pandemic periods [9]. If deemed necessary sensitivity analysis adding 'pandemic enrolment period' into the model will be run and if found to be significant subgroup analysis may be conducted.

Finally, as indicated in section 4.6 an evaluation of missing data will be conducted prior to analysis. Missing data will be assessed by 'pandemic enrolment period' to check whether there are any differences of missingness caused by the pandemic. Missing data will be handled in line with section 4.6 of this SAP with additional guidance from recent literature on dealing with missing data in a pandemic [10].

One element of study processes which have been largely impacted by COVID is the data collection of the UDS, which will have an impact on the primary outcome. Essentially this is seen as missing data but it doesn't impact the level of missing data just the reliability of the self-report and occurs in both arms of the trial. The trial originally planned to collect UDS tests every two weeks however the following occurred;

Table 3: Summary of UDS data collection during trial following COVID-19 impacts

| Site | Date | UDS dat | a collection |
|------|----------------------------------|---------------|-------------------|
| | | TAU arm | Intervention arms |
| All | Up to 2 <sup>nd</sup> April 2020 | every 2 weeks | every 2 weeks |

| All | 2 <sup>Nd</sup> April 2020 – 12 <sup>th</sup> June | Not collected | Not collected |
|---|---|---|---|
| | 2020 | | |
| South London | 04.05.2020 | Not Collected | Monthly |
| | 12.06.20 | Monthly | Monthly |
| Newcastle | 07.05.2020 | Not Collected | Monthly |
| | 29.06.20 | Monthly | Monthly |
| Manchester | 13.07.20 | Monthly | Monthly |
| West Midlands | 03.07.20 | Monthly | Monthly |
| Tayside opened for | 27.07.20 | Monthly | Monthly |
| recruitment on | is . | | |

As at the point of writing the SAP the trial is continuing to collect UDS monthly (on the larger visit weeks 4,8, 12, 16,20, 24). As there is little study data that hasn't been impacted by this and it has affected both arms simultaneously sensitivity analysis around this is not required. If any further changes during the ongoing pandemic occur that the investigators feel will impact any signal detected this will be conducted as exploratory post-hoc analysis.

### **6.10 EXPLORATORY ANALYSES**

As indicated in section 5.2, further analysis is to be conducted at a later date but will not form the results of the current analysis. A separate statistical plan detailing all other analysis will be written and published in addition to this SAP.

### 7. SOFTWARE

All quantitative analysis will be completed using STATA version 15 or later.

# 8. REFERENCES

- Peacock A et al. Global statistics on alcohol, tobacco and illicit drug use: 2017 status report. Addiction. 2018 May 10. doi: 10.1111/add.14234.
- 2. White, I. R., Royston, P., & Wood, A. M. (2011). Multiple imputation using chained equations: issues and guidance for practice. Statistics in medicine, 30(4), 377-399.

- 4. Sobell L. C., Sobell M. C., Leo G. I., Cancilla A. Behavioral assessment and treatment planning with alcohol and drug abusers: a review with emphasis on clinical application. *Clin Psych Rev* 1988; 8: 19–54.
- 5. Fals-Stewart W., O'Farrell T. J., Freitas T. T., McFarlin S. K., Rutigliano P. The timeline followback reports of psychoactive substance use by drug-abusing patients: psychometric properties. *J Consult Clin Psychol* 2000; **68**: 134–44.
- 6. Sobell, Linda & Sobell, Mark. (1992). Timeline follow-back: A technique for assessing self-reported alcohol consumption. Measuring Alcohol Consumption: Psychosocial and Biochemical Methods. 41-72.
- 7. Grubbs, F. E. (1969). Procedures for detecting outlying observations in samples. Technometrics, 11(1), 1-21.
- 8. See: <a href="https://www.gov.uk/government/publications/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-commissioners-and-providers-of-services-for-people-who-use-drugs-or-alcohol/covid-19-guidance-for-pe
- 9. Meyer et al (2020): Statistical Issues and Recommendations for Clinical Trials Conducted During the COVID-19 Pandemic, Statistics in Biopharmaceutical Research, DOI: 10.1080/19466315.2020.1779122
- 10. Cro, S., Morris, T.P., Kahan, B.C. et al. A four-step strategy for handling missing outcome data in randomised trials affected by a pandemic. BMC Med Res Methodol 20, 208 (2020). https://doi.org/10.1186/s12874-020-01089-6

### **APPENDICES**

APPENDIX 1 - POISSON REGRESSION ANALYSIS DECISION TREE

APPENDIX 2 – OBJECTIVES AND ASSOCIATED OUTCOME MEASURES AND CHARACTERISTICS

APPENDIX 3 - OUTCOME MEASURES SUMMARY AND SCORING TABLE

APPENDIX 4 - ASSUMPTIONS OF MODELS

### APPENDIX 1 - POISSON REGRESSION ANALYSIS DECISION TREE



Figure obtained from;

https://pdfs.semanticscholar.org/8ab1/829f559b869eeb48e38f15c5d94dc957a0f5.pdf

APPENDIX 2 – OBJECTIVES AND ASSOCIATED OUTCOME MEASURES AND CHARACTERISTICS

| Objective | Outcome Measure | Time Period | End point | Variable<br>Type | Analysis<br>Model | Scoring |
|---|---|---|---|---|---|---|
| One - effectiveness of | Primary outcome | | | | | |
| BUP-XR and MET/BUP-<br>SL | Number of days abstinent from heroin | Days 8 – 168 | 24 weeks | Count | Poisson<br>Regression | Count of days abstinent |
| | Secondary outcomes | | | | | |
| | Number of days abstinent from cocaine | Days 8 – 168 | 24 weeks | Count | Poisson<br>Regression | Count of days abstinent |
| | Number of days abstinent from<br>Benzodiazepines | Days 8 – 168 | 24 weeks | Count | Poisson<br>Regression | Count of days abstinent |
| | Longest time in days continuously abstinent from heroin | Days 8 – 168 | 24 weeks | Count | Poisson<br>Regression | Max Count of days consecutively abstinent |
| | Longest time in days continuously abstinent from cocaine | Days 8 – 168 | 24 weeks | Count | Poisson<br>Regression | Max Count of days consecutively abstinent |
| | Longest time in days continuously abstinent from Benzodiazepines | Days 8 – 168 | 24 weeks | Count | Poisson<br>Regression | Max Count of days consecutively abstinent |
| Two – Safety profile | Number of safety events | Study enrolment to 24 weeks | 24 weeks | Count | Descriptive | n/a |
| Three – Treatment<br>retention | Total retention time | Days 8 – 168 | 24 weeks | Count | Poisson<br>Regression | Count of Days enrolled in maintenance medication for OUD |
| | Survival time to study withdrawal | Randomisation date to first discontinuation | 24 weeks | Time to event | Cox<br>regression | Time to first discontinuation |
| Four – OUD and CUD remission status | SCID-RV interview | Baseline to week 24 | 12 weeks & 24<br>weeks | binary | (Binary)<br>logistic | Remission status (Yes/No) indicated by SCID-RV (see |
| | ā | | 8 5 | | regression | appendix 3 for SCID scoring) |

# APPENDIX 3 - OUTCOME MEASURES SUMMARY AND SCORING TABLE

| Standard Clinical interview for Dependence — Research version SCID-RV No reference available; below scoring derived from MACRO database | | | 65 | | ealles | |
|---|---|---|---|---|---|---|
| No reference available; below scoring d | ance - Research version SCID-R | <b>A</b> | | | | |
| | lerived from MACRO database | | | | | |
| Structured Clinical Interview for Two single item scales (one for | single item scales (one for | Items are coded on a 5 point | None found | Lower better | None found | None found |
| DSM-5 (SCID-5) is a semi opioi | opioid and one for cocaine). | scale based on number of | | | | |
| structured interview guide for | 2 | symptoms present; | | 20 | | |
| making the major DSM-5 Remi | Remission status is to be | Œ | | | | |
| diagnoses. calcu | calculated from the SCID. | no symptoms, 1 symptom, | | | | |
| Rem | Remission is satisfied (i.e. 'yes') if | Mild (2 – 3), Moderate (4-5) | | | | |
| (s ou | no symptoms are present that is a | and Severe (6 or more) | | 8 | | 28 |
| score | score of 1 or lower is obtained. If | | 20 | | 00 | |
| a scc | a score of 2 or more is given then | | | | | 5 |
| remi | remission status is 'no'. | | | | | |
| Clinical Global Impression scale (severity and improvement - CGI-S/CGI-I) | ty and improvement - CGI-S/CG | (1-1) | | | | |
| Busner, J. and Targum, S.D., The Clinical Global Impressions Scale: Applying a Research Tool in Clinical Practice (2007). Psychiatry. | I Global Impressions Scale: App | lying a Research Tool in Clinical F | ractice (2007). Psychiatry. | | | |
| Brief stand-alone Two | Two single item scales (CGI-S and | The CGI severity ranges | 1. Severity (1 | Lower better | None found | 1 – Extremely mild |
| assessment of the clinician's GCI-I | GCI-I). Both items individually | from 1 'extremely mild' to | item) | 1 | ; | 2-Very mild |
| view | scored on a 1 to 7 point scale. | 7 'extremely severe' | 550 | | | 3 – Mild |
| of the patient's global | | 20 | | | | 4 – Moderately severe |
| functioning. The scale Total | Total score is not to be calculated | | | | 25 | 5 – Severe |
| comprises two from | from the two scales. However, | 8 | E 8 | 70 | | 6 – Very severe |
| companion one-item measures the t | the two scale scores will range | | | 89 | | 7 – Extremely severe |
| evaluating the from | from 1 to 7. | The CGI improvement | 2. Improvement | Lower better | | 1- very much improved |
| severity of psychopathology | | ranges from 1 'very much | (1 item) | 300 | 11 | 2 – much improved |
| and change from the | | improved' to 7 'very much | | 3 | | 3 – minimally improved |
| initiation of treatment. | - 28 | worse' | | | | 4 – no change |
| | ž. | | | | | 5 – minimally worse |
| 8 | 34<br>34 | | | T . | | 6 – much worse |
| | | ± 00 | | | 8 8 | 7 – very much worse |

| Used for substance use | A 14 item measure consisting of | Items 1, 3, 4, 5, 9, 10 rated; | 1. Addiction severity | 1. Higher scores indicate | None found | 1. Low 0 – 1, moderate |
|---|---|---|---|---|---|---|
| SUD) clinicians | | 0 'None' and 1 'Present' | (items $1-3$ ). | worse | | 2-3 and high 5-4 |
| obtain a brief multi dimension<br>patient profile of addiction<br>related severity, health and | | Items 2, 5, 6, 7, 8, 11, 12, 13, 14 rated 0 'None', 1 'Low', 2 | Coexisting problem complexity (items 4 – 10) | 2. Higher scores indicate better | | 2. Low 0 – 2, moderate<br>3 – 5 and high 6 – 15 |
| social problem complexity and recovery strengths | in the subscale. | Modelate allo mall. | 3. Recovery Strengths | 3. Higher scores indicate | | 3. Low 0 – 5, moderate |
| | An overall measure total score is not obtainable, just 3 subscale | 8 | (items 11 – 14) | better | | 6 – 8 and high 9 – 11 |
| | scores. | ū | ٠ | (A) | | |
| 18 | 1. total range 0 – 5 | 8 | | = | | 12 |
| 27 | | | | 2000 | | |
| | <ol> <li>total range U − 11</li> </ol> | | | | | |
| Craving response using Craving 6 | Craving response using Craving experience questionnaire (CEQ-F) | | | | | |
| No reference available; below sc | No reference available; below scoring derived from MACRO database | | | | | |
| Craving Experience | 11 item scale. | Each item rated on a scale | None identified | indicate more | None found | None found |
| Questionnaire | | from 0 – 10. | | severe craving | | |
| 5 | Total scale calculated by | | | 5 | | |
| | summing the 11 items, therefore | | | | | #I |
| | final score ranges from 0 to 110. | | | B 9 | | |
| Visual analogue craving rating (Need/Want) (VAS-N/VAS-W) | Veed/Want) (VAS-N/VAS-W) | | | | | |
| No reference available; below sc | No reference available; below scoring derived from MACRO database | | | | | |
| Self-report craving rating | Two individual items one | Both items are scored on a 0 | None identified | Higher scores indicate more | None found | None found |
| | measures rating need and the | - 100 continuous scale | | severe craving | | |
| | other rating want. | | | 60 | | |
| | | 28 | | 5 | | |
| | Total score is not to be calculated | | | | | - N |
| nt (2) (3) | from the two scales. However, | | | 8 | | |
| W | the two scale scores will range | 18 | | | | |
| | from 0 to 100. | 2 | 22 | | | |
| | 3 | | | | | |
| Social functioning using Work ar | Social functioning using Work and Social Adjustment Scale (WSAS) | | | | | |
| Mundt, J.C., et al., The Work and | Mundt, J.C., et al., The Work and Social Adjustment Scale: a simple measure of impairment in functioning (2002). British Journal of Psychiatry, 180, 461 – 464 | easure of impairment in function | ning (2002). British Journal o | f Psychiatry, 180, 461 – 464. | | 上 先生 新作品 水流 医 · |

Page | 41

| 42 |
|------|
| Page |

| Self-report scale of functional | Five item scale. Total score | Items rated on a 0 to 8 scale | None identified | Higher scores indicate better | None found | None found |
|---|---|---|---|---|---|---|
| impairment attributable to an | calculated by summing up 5 items | with 0 indicating no | | state. | | |
| identified problem. | in the scale. | impairment and 8 indicating | | | | |
| 25 | ^ | very severe impairment | | | | |
| | Total score ranges from 0 - 40 | | | | | |
| Quick inventory of Depressive Symptomatology (QIDS-SR) | mptomatology (QIDS-SR) | | | | | |
| Rush, A. J., Trivedi, M. H., Ibrahin | Rush, A. J., Trivedi, M. H., Ibrahim, H. M., Carmody, T. J., Arnow, B., Klein, D. K., Keller, M. B. (2003). The 16-Item quick inventory of depressive symptomatology (QIDS), clinician rating (QIDS-C), and self- | sin, D. K., Keller, M. B. (2003). | The 16-Item quick inventory | / of depressive symptomatology ( | (QIDS), clinician ra | ting (QIDS-C), and self- |
| report (QIDS-SR): a psychoMETric | report (QIDS-SR): a psychoMETric evaluation in patients with chronic major depression. Biological Psychiatry, 54, 573-583 | najor depression. Biological Psy | chiatry, 54, 573-583. | | | |
| self-report measure of | self-report measure of 16 item scale. | Items rated on a 0 to 3 scale: | 1 Sleen distrirbance | Higher scores worse for all | None found | For total score |
| | | O indicating no symptom and | (items 1 | subscales | | |
| | Subscales calculated by taking | 3 indicating worse. | 2. Sad mood (item 5) | | | 1-5 = No depression |
| 5 | highest score of any one item of | | 3. Decrease/increase | | | 6-10 = Mild depression |
| | the subscale. Total score for each | * | | 2 8 | | 11-15 = Moderate |
| 6 | subscale ranging from 0 to 3 | | weight (items 6 - 9) | | | depression |
| 5 | | | 4. Concentration | | | 16-20 = Severe |
| | Total score calculated by | | (item 10) | | | depression |
| a a | summing the 9 subscales | | 5. Self-criticism (item | | | 21-27 = Very severe |
| | therefore total scores range from | | 11) | | | depression |
| | 0 to 27. | | 6. Suicidal ideation | | | |
| - t/2 | 2 | 6) | (item 12) | | | |
| | | | 7. Interest (item 13) | | | |
| 8. | . 8 | | 8. Energy/fatigue | | | |
| | 2 | | 9. Psychomotor | | | |
| | 2 | | | | | |
| | 100 | | retardation (items | | | = |
| Improvement and Recovery using | Improvement and Recovery using Substance Use Recovery Elevator (SURE) | URE) | | | | |
| Neale, J., Vitoratou, S., Finch, E., I | Neale, J., Vitoratou, S., Finch, E., Lennon, P., Mitcheson, L., Panebianco, D., Rose, D., Strang, J., Wykes, T., Marsden, J. (2016) 'Development and validation of 'SURE': A patient | o, D., Rose, D., Strang, J., Wykes, | T., Marsden, J. (2016) 'Deve | elopment and validation of 'SURE | ': A patient | |
| reported outcome measure (PRO | reported outcome measure (PROM) for recovery from drug and alcohol dependence', | ol dependence', Drug and Alcoh | ol Dependence. DOI: 10.101 | , Drug and Alcohol Dependence. DOI: 10.1016/j.drugalcdep.2016.06.006 | | |
| Self-report measure to assess | 21 item scale. | Section A (items 1 – 3) rated | 1. Drinking and drug | Individual items indicates | None Found | None Found |
| person al recovery from drug | = | | use (items 1 – 6) | lower better and higher | | |
| and/or alcohol dependence | Items 1 – 3 scored; | ranging from 1 'Never' to 5 | 2. Self-care (items 7 – | worse but scores are then | | 100 Miles |
| | | evelyday | 11) | weighted higher if lower so | | |

| 3 | Wever' OR 'On 1 or 2 days' = $3$ , | | <ol><li>Relationships</li></ol> | total score tormat is higher | | |
|---|---|---|---|---|---|---|
| | And Back to act | Section B (items 7 - 21) | (items 12-15) | correc indicate hetter | | |
| lise s | Oil 3 Oil 4 days = 2, Oil 3 Oil 9 | _ | (CT TT CILITY) | | _ | , |
| 80 | days' OR 'Every day' = 1 | rated on a 5-point scale I - | Rankerial | | | 0 2 |
| | | 5; ranging from 1 'none of | 4. Material resources | | 903 | |
| _ | Items 4 – 21 scored; | the time' to 5 'all of the | (items 16 – 18) | | 8 | |
| | 'All of the time' OB 'Most of the | time'. | 100 | 307 | 22 | |
| | THE PROPERTY OF THE PARTY OF TH | | S. Outlook on line | | | |
| | time = 3, A rair amount of the | Soution Citame and used for | (items $19 - 21$ ) | | | |
| | time' = 2, 'A little of the time' UR | _ | | | | _ |
| | 'None of the time' = 1 | measure scoring. | | 级 | | |
| 2 | | | | | | N |
| 7 | Score range for each subscale | 8 | | | | |
| | R | -20 | | 2 | | |
| | Orinking and drug 180. 6.1.18 | | | | | |
| 1 | | | | <b>V</b> | , | |
| | 2. Self care; 5 – 15 | lu | | | 2 | 8 |
| × | 3. Relationships; 4 – 12 | | | | | |
| 29 | 4. Material resources: 3 – 9 | | | | | 9 |
| W | | 20 | | | | 6 |
| 8 | | | | | | |
| | Total score ranges from 21 – 63 | | | | | |
| Patient Reported Outcome State | Patient Reported Outcome Status (severity and improvement - PRO-S/PRO-I) | S/PRO-I) | | | | |
| No reference available; below su | No reference available; below scoring derived from MACRO database | | | | | |
| Patient reported outcome of | Two single item scales (PRO-S | The PRO severity ranges | 1. Severity (1 item) | Lower better | None found | 1 – Extremely mild |
| severity and improvement of | and PRO-I). Both items | from 1 'extremely mild' to | | | | 2-Very mild |
| addition problem | individually scored on a 1 to 7 | 7 'extremely severe' | | 0 | | 3 – mild |
| , | point scale. | | | 5 | 3 | 4 – moderate |
| | 8 | | | | | 5 - severe |
| 40 | Total score is not to be calculated | 81 100 | | | | 6 – very severe |
| 0 | from the two scales. However, | 8 | | x | 14 | 7 – extremely severe |
| 19 | the two scale scores will range | The PRO improvement | 2. Improvement (1 | Lower better | a | 1-very much improved |
| | from 1 to 7. | ranges from 1 'very much | item) | | | 2 - much improved |
| | | improved' to 7 'very much | | | ** <sub>0</sub> | 3 – minimally improved |
| | | worse' | | 2 | s | 4 – no change |
| | | | | II | | 5 - minimally worse |
| | | | | 1)<br>3) | | 6 – much worse |
| | | 4 | | | je<br>M | 7 - very much worse |
| Emotion regulation using the Di | Emotion regulation using the Difficulties in Emotion Regulation Scale- short form (Emotion regulation using the Difficulties in Emotion Regulation Scale- short form (DERS-SF) | - short form (Emotion regulation | using the Difficulties in Em | stion Regulation Scale- short for | n (DERS-SF)) | |
| | | | | | | 3 |

| 44 |
|------|
| Page |

| | | , | | | Million English | N 1 C |
|---|---|---|---|---|---|---|
| self-report measure for | 18 item scale | ıŋ | 1. Strategies (items | Lower scores indicate better | None tound | None round |
| assessing emotion regulation | Items in each scale summed to | point scale ranging from 1 | 10, 15 and 18) | | | |
| problems | give individual scale scores | Never' to 5 'Almost | 2. Non-acceptance | awareness scale (items 1, 4 | | |
| | (ranging from 1 to 5) and total | always′ | (items 7, 12 and 16) | and 6) lower scores indicate | , | |
| | score calculated by summing | Awareness snale should be | 3. Impulse (items 9, 14 | worse | | |
| | scales, total score ranging from 18 | | and 17 | × | | • |
| | to 90 | | 4. Goals (items 8, 11 | | | |
| ű. | Đ | to 5 'almost never'. | and 13) | St. | | |
| | | | 5. Awareness (items 1, | | 117 | |
| | 19. | 2 | 4 and 6) | | | |
| | | 9 | 6. Clarity (items 2, 3 | | | |
| ě | | | and 5) | 2 | | |
| Alcohol quantity, frequency, max | Alcohol quantity, frequency, maximum consumption (ALC-QF (TOP)) | | | | | |
| No reference available; below sco | No reference available; below scoring derived from MACRO database | | | | | |
| Alcohol – typical Quantity and | 3 items in measure; number of | Items rated based on N | None found | Higher numbers indicate | None found | None found |
| Frequency. Using an adapted | days, average units and maximum | number of drinking days in | | more drinking days and units. | | |
| version of the Treatment | units on any given day. | past four weeks; 0 to 28 | 12 | | | |
| Outcomes Profile (TOP). The | | | | | | 98 |
| TOP is the standard national | Maximum units will be reported | Units given on scale from 0 | | | | ñ |
| instrument for monitoring the | descriptively. Quantity and | to 100 | | ū | | |
| outcomes of public substance | Frequency will be treated as two | | | | | |
| use disorder treatment services | separate items. | Maximum units ranges from | | | | |
| in England. | | 0 to 500. | | | | |
| The Montreal Cognitive Assessment (MoCA) | ent (MoCA) | | | | | |
| Original ref: Nasreddine Z.S., Phil | Original ref: Nasreddine Z.S., Phillips N.A., Bédirian V., Charbonneau S., Whitehead | , Whitehead V., Collin I., Cumming | gs JL, Chertkow H. The Mo | V., Collin I., Cummings JL, Chertkow H. The Montreal Cognitive Assessment (MoCA): A Brief Screening Tool for Mild Cognitive | CA): A Brief Screen | ing Tool for Mild Cognitive |
| Impairment, Journal of the Amer | mpairment, Journal of the American Geriatrics Society. 53 (2005) 695-699. | -699. | | | | |
| Evaluates whether someone's | 10 Item scale, with an additional | 10 items are rated on N | None found | Higher numbers indicate less | If Item 11 | A score of 26 or above is |
| thinking ability is impaired | item (No. 11) to indicate | various scales (0 to 1, 2, 3, 5 | 400 | cognitive impairment | (education | considered normal. |
| | education level. | and 6) | | , | level) is missing | |
| ¥ | tems 1-10 are summed together | 25 | | | should still be | |
| 2 | to give a total score ranging from | | | × | calculated. | O.Ba |
| | 0 to 30. | • | | | | |
| | | | 90 | | | |

| | N | | 22 |
|---|---|---|---|
| 8 | | | |
| | 26 | | |
| | | æ | <br>A <sub>111</sub> |
| 2 | | | |
| | , | | |
| | 1 9 | | |

An extra point is awarded if item 11 is 'Yes' (i.e. subject has 12 years or fewer of formal However, the max score is 30 so If a participant scores 30 out of 30 this additional point isn't added.

education),

# **APPENDIX 4 – ASSUMPTIONS OF MODELS**

| Assumption | Checking |
|---|---|
| Poisson Regre | ession |
| distribution of counts (conditional on the model) follow a | calculate the expected counts and plot these with |
| Poisson distribution | the observed counts to see if they are similar |
| The mean and variance of the model are identical | Graphical display |
| | Pearson dispersion statistic |
| If you satisfy this assumption you have equidispersion. | |
| often this is not the case and your data are either under- | See appendix 1 for more detail. |
| or over dispersed. | see appendix 2 for more detain |
| Generalised Linear | nived model |
| Linearity | scatter plots of the model residuals vs predictor |
| Linearity | scatter plots of the model residuals vs predictor |
| the relationship between the independent and | |
| dependent variables to be linear | |
| U8Residuals/errors are independent | Scatter plot |
| Obkesiduais/errors are independent | Durbin-Watson test |
| Little on the completion in the date (special release beauty) | Durbin-watson test |
| Little or no autocorrelation in the data. (residuals should | |
| be independent from each other) | |
| Residuals/Errors are normally distributed | Q-Q-Plot |
| Residuals/Errors have constant variance | Scatter plot of standardized residuals versus |
| | predicted values |
| There should be no homoscedasticity of error terms | |
| No or little multi-collinearity | inspection of correlation coefficients and |
| | Tolerance/VIF values |
| (independent variables should not be highly correlated | |
| with each other) | |
| ORDINAL LOGISTIC | REGRESSION |
| There should be no multi-collinearity | inspection of correlation coefficients and |
| | Tolerance/VIF values |
| You should have proportional odds | full likelihood ratio test comparing the fit of the |
| | proportional odds model to a model with varying |
| | location parameters |
| BINARY LOGISIC R | EGRESSION |
| Linear relationship between the continuous independent | Box-Tidwell (1962) procedure |
| variables and the logit transformation of the dependent | 2 |
| variable. | # S |
| Your data must not show multi-collinearity | inspection of correlation coefficients and |
| | Tolerance/VIF values |
| There should be no significant outliers, high leverage | Box plots |
| points or highly influential points | BOX PIOUS |
| Cox regression | n model |
| proportional hazards | Kaplan Meier curves |
| proportional nazards | Napidii Micici Cui Ves |
| the ratio of the hazards for any two individuals is | |
| | 4 |
| constant over time | |
| linear covariate relationships | residual plots |
| The Cox model assumes that each variable makes a linear | |
| contribution to the model | |